CLINICAL TRIAL: NCT06807255
Title: Lactate Values During Labour and Their Correlation With Maternal and Foetal Outcome: a Prospective Observational Single-centre Study
Brief Title: Lactate Values During Labour and Their Correlation With Maternal and Foetal Outcome
Status: Completed | Type: Observational
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Barbara Milan, MD, Papa Giovanni XXIII Hospital
Other Study IDs: REF: no. 751/2023, reg56/23
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Lactate Values During Labour in Women Receiving Neuraxial Anaesthesia
Keywords: Lactate values during labour,; maternal and foetal outcome; HIFI; myometrial contraction; lactacidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lactate levels were assessed via a venous blood gas test utilising an IV cannula already placed in the woman's limb upon admission — Lactate levels were assessed via a venous blood gas test utilising an IV cannula already placed in the woman's limb upon admission; subsequent analysis was conducted using rapid processing (under 5 minutes from the pre-test) with the Rapidpoint 500 Systems-Siemens (Siemens, Milano) emogasanalyzer

SUMMARY:
Postpartum haemorrhage (PPH) represents a significant cause of morbidity in the obstetric population, with a mortality rate of 140,000 women per year, and the predominant cause of PPH (70%) is uterine atony.

Consequently, elevated lactate levels during labour could influence maternal and foetal well-being. We decided to assess lactate concentrations during labour in women receiving neuraxial anaesthesia and evaluate the association between high lactate levels and adverse maternal and foetal outcomes.

The secondary aims of the study were to assess lactate levels at different stages of labour and investigate whether increased lactate concentrations could influence neonatal cord pH upon delivery.

DETAILED DESCRIPTION:
We conducted a prospective observational single-centre study involving women in active labour receiving neuraxial anaesthesia.

Labour analgesia was placed at the beginning of active labour, whose definition follows the NICE guidelines. The labour analgesia technique consisted of standard epidural puncture or dural puncture epidural; the maintenance of analgesia was through clinician intermittent boluses given on maternal request.

Lactate levels were assessed via a venous blood gas test utilising an IV cannula already placed in the woman's limb upon admission.

These measurements were taken at three different time points, as follows: T0: at the time of diagnosis of the active phase of the first stage of labour, T1: at the beginning of the active phase of the second stage of labour, at the beginning of active pushing, and T2: at the time of the delivery, before placenta expulsion.

Postpartum haemorrhage (PPH) has been defined following the definition of the Royal College of Obstetricians and Gynaecologists as a total blood loss ≥ 500 ml.

To measure umbilical cord pH, 1-2 ml of cord blood were taken from the umbilical artery one minute after birth, regardless of clamping.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* single pregnancy with a gestational age of ≥ 36 weeks
* active labour with a cervix dilation of 4 to 6 cm
* neuraxial analgesia
* consent to the study Exclusion criteria
* < 18 years
* twin pregnancy
* gestational age < 36 weeks,
* labour without labour analgesia
* cervix dilation > 6 cm at the moment of the placement of neuraxial analgesia
* not consent to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: women in active labour receiving neuraxial anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
the primary aim of our study was to assess whether elevated lactate values during labour are associated with an increased risk of PPH | two hours
  Postpartum haemorrhage has been defined following the definition of the Royal College of Obstetricians and Gynaecologists as a total blood loss ≥ 500 ml.
  Our population was divided into two groups: those with total blood loss ≤ 500 ml and those with blood loss > 500 ml.

SECONDARY OUTCOMES:
The secondary aims of the study were to assess lactate levels at different stages of labour and investigate whether increased lactate concentrations could influence neonatal cord pH upon delivery | Time of labour
  Measurements were taken at three different time points, as follows: T0: at the time of diagnosis of the active phase of the first stage of labour, T1: at the beginning of the active phase of the second stage of labour, at the beginning of active pushing, and T2: at the time of the delivery, before placenta expulsion.
neonatal cord pH upon delivery | five minutes
  To measure umbilical cord pH, 1-2 ml of cord blood were taken from the umbilical artery one minute after birth, regardless of clamping.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Fierro, MD, Study Chair — ASST Papa Giovanni XXIII
Locations (1):
- ASST Papa Giovanni XXIII, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: Yes
If requested by the reviewer, it will be possible to share the anonymised database
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 29/01/2025 for ten years
Access Criteria: If requested by the reviewer, it will be possible to share the anonymised database

REFERENCES:
- [Background] Prevention and Management of Postpartum Haemorrhage: Green-top Guideline No. 52. BJOG. 2017 Apr;124(5):e106-e149. doi: 10.1111/1471-0528.14178. Epub 2016 Dec 16. No abstract available. PMID 27981719
- [Background] Alotaibi M, Arrowsmith S, Wray S. Hypoxia-induced force increase (HIFI) is a novel mechanism underlying the strengthening of labor contractions, produced by hypoxic stresses. Proc Natl Acad Sci U S A. 2015 Aug 4;112(31):9763-8. doi: 10.1073/pnas.1503497112. Epub 2015 Jul 20. PMID 26195731
- [Background] Hanley JA, Weeks A, Wray S. Physiological increases in lactate inhibit intracellular calcium transients, acidify myocytes and decrease force in term pregnant rat myometrium. J Physiol. 2015 Oct 15;593(20):4603-14. doi: 10.1113/JP270631. Epub 2015 Sep 3. PMID 26223765